CLINICAL TRIAL: NCT04994223
Title: Effectiveness of Combined Anticoagulation and Antithrombotic Therapy vs Antithrombotic Therapy Alone After Lower Extremity Revascularization for Peripheral Arterial Disease
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Armed Forces Post Graduate Medical Institute (AFPGMI), Rawalpindi (Other)
Responsible Party: Principal Investigator, Ayesha Masood, Trainee in vascular surgery, Armed Forces Post Graduate Medical Institute (AFPGMI), Rawalpindi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PAD
Record Dates: First submitted 2021-07-30; First posted 2021-08-06 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Combined Anticoagulation and Antithrombotic Therapy; PAD - Peripheral Arterial Disease
Keywords: rivaroxaban in PAD
MeSH Terms: interventions — Rivaroxaban; Tablets

STUDY DESIGN:
Intervention Model Description: patients enrolled in the study would be taken informed consent and divided in two groups, group A receiving rivaroxaban plus aspirin and Group B receiving placebo plus aspirin
Who Masked: Participant, Investigator
Masking Description: participants enrolled in the study and the principal investigator would not be knowing the drug regimens used in group A and Group B participants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A(combined anticoagulation plus antithrombotic therapy group) (Experimental): group A patients would be receiving rivaroxaban and aspirin as experimental group to see the efficacy of rivaroxaban in peripheral arterial disease.
  Interventions: Drug: Rivaroxaban 10 MG Oral Tablet [Xarelto]
- Group B( antithrombotic therapy alone group) (Active Comparator): group B patients would be those receiving traditional antithrombotic therapy as usually given n Peripheral Arterial Disease.
  Interventions: Drug: Rivaroxaban 10 MG Oral Tablet [Xarelto]

INTERVENTIONS:
Drug: Rivaroxaban 10 MG Oral Tablet [Xarelto] — rivaroxaban has shown improved results after revascularization for PAD in terms of limb survival

SUMMARY:
EFFECTIVENESS OF COMBINED ANTICOAGULATION AND ANTITHROMBOTIC THERAPY VS ANTITHROMBOTIC THERAPY ALONE AFTER LOWER EXTREMITY REVASCULARIZATION FOR PERIPHERAL ARTERIAL DISEASE.

DETAILED DESCRIPTION:
Anticoagulation and antithrombotic therapy is a crucial part of PAD management as it prolongs the patecy of grafts in open surgical revascularization procedures so its proper dosage and duration without increasing risks to the patient and maximizing the benefits is very important.

Currently literature in Pakistan regarding this problem couldn't be found so this study would help assessing the outcomes of anticoagulation and antithrombotic therapy in this population with respect to treatment options available and presentation variability of the peripheral arterial disease. Patients with PAD would be enrolled for 6 months and would be followed upto 12 months and then upto 24 months.

Eligible subjects will be randomized 1:1 to receive either rivaroxaban 5 mg twice daily plus aspirin 75 mg once daily or rivaroxaban-matching placebo twice daily plus aspirin 75 mg once daily stratified by type of procedure; the treatment assignment will be double-blinded. Randomization and study treatment will begin as soon as possible but no later than 10 days after a successfull lower extremity revascularization.

Patients will be prohibited from taking any additional antithrombotic therapy other drugs, including anticoagulants, doses of aspirin >100 mg daily, vorapaxar, ticagrelor, prasugrel, or cilostazol. Enrolled subjects will be having symptomatic PAD defined by evidence of an abnormal ankle-brachial index ≤0.80 in either limb with an anatomy of occlusive disease of involving segments. Subjects would be randomized who had undergone a technically successful endovascular, hybrid, or surgical LER within 10 days and had achieved adequate hemostasis before randomization.

ELIGIBILITY:
Inclusion Criteria:

- all patients with PAD candidates for revascularization procedures

Exclusion Criteria:

1. planned long-term dual antiplatelet therapy (>6 months),
2. clinical requirement for therapeutic anticoagulation,
3. recent acute limb ischemia or acute coronary syndrome,
4. medical condition that could increase the risk of major bleeding, significantly impaired renal function at baseline (estimated glomerular filtration rate <15 mL•min-1•1.73 m-2),
5. any documented history of intracranial hemorrhage, stroke, or transient ischemic attack

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-07-02 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
ALI | upto 1 year
  acute limb ischemia
major amputation for vascular reasons | upto 1 year
  any type of major amputation after revascularivation for PAD
MI | upto 1 year
  myocardial infarction
ischemic stroke | upto 1 year
  ischemic stroke
cardiovascular death | upto 1 year
  death because of cardiovascular events

SECONDARY OUTCOMES:
thrombolysis in myocardial infarction(TIMI)major bleeding | 2, 30, 180 and 365 days
  combined therapy effect may result in increased bleeding tendency

CONTACTS AND LOCATIONS:
Locations (1):
- Combined Military Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
title
Supporting Information: Study Protocol
Time Frame: 6 months from start of study